CLINICAL TRIAL: NCT02060812
Title: The Effect of Sono-guided Suprascapular Nerve Block Combined With Axillary Nerve Block in Arthroscopic Rotator Cuff Repair: a Randomized Controlled Trial
Brief Title: Axillary Nerve Block Combined With Suprascapular Nerve Block
Acronym: SSNBANB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Assistant professor in department of orthopedic surgery, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSNB&ANB; Chuncheon1 (Other: Chuncheon)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Rotator Cuff Tear
Keywords: ultrasound guided axillary nerve block; arthroscopic rotator cuff repair; ultrasound guided suprascapular nerve block; rebound phenomenon of pain
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I, SSNB & ANB (Experimental): 21 patients were randomly allocated into group I, and received suprascapular nerve block (SSNB) and axillary nerve block (ANB) both with 10mL ropivacaine.
  Interventions: Procedure: Group I, SSNB & ANB
- Group II, SSNB alone (Placebo Comparator): The other 21 patients were allocated into group II, and received suprascapular nerve block (SSNB) with 10mL ropivacaine and axillary nerve block (ANB) with placebo (10mL normal saline).
  Interventions: Procedure: Group II, SSNB alone

INTERVENTIONS:
Procedure: Group I, SSNB & ANB — Suprascapular nerve block (SSNB) and axillary nerve block(ANB) were performed by one anesthesiologist under sono-guidance. 23 gauge spinal needle was used. SSNB was done at first and the entry site was the mid point between an anterolateral angle of acromion and medial end of scapular spine. With the linear probe, the suprascapular notch was identified and the block was performed penetrating the transverse scapular ligament because the scapular nerve and artery were located at the suprascapular notch. Just after the SSNB, ANB was performed and the entry site was the point 1.5 cm medial and 2cm inferior to posterolateral angle of acromion. With the linear probe, posterior circumflex artery was identified and the block was done at just above the artery.
  Arms: Group I, SSNB & ANB
Procedure: Group II, SSNB alone — This is same as the Group I, SSNB & ANB, but ANB was performed with placebo(10mL normal saline).
  Arms: Group II, SSNB alone

SUMMARY:
Purpose: The purpose of this study is to compare the result of combined sono-guided suprascapular nerve block (SSNB) and axillary nerve block (ANB) with isolated SSNB in postoperative pain following arthroscopic rotator cuff repair. Our hypothesis was that SSNB combined ANB would show a more effective anesthesia for arthroscopic rotator cuff repair as compared with SSNB only.

Methods: Forty-two patients with rotator cuff tear who had undergone arthroscopic rotator cuff repair were enrolled in this study. Among them, 21 patients were randomly allocated into group I, and received SSNB and ANB with each 10mL ropivacaine. The other 21 patients were allocated into group II, and received SSNB with 10mL ropivacaine and ANB with 10mL normal saline. Visual Analogue Scale (VAS) pain score, patient's satisfaction (SAT), and Lateral Pain Index (LPI), etc was checked at postoperative 1, 3, 6, 12, 18, 24, 36, and 48 hours.

DETAILED DESCRIPTION:
All procedures described in the present study were approved by the Institutional Review Board of our hospital, and all patients gave written informed consent to participate in the present study. Between November 2012 and July 2013, forty-two patients with rotator cuff tear who had undergone arthroscopic rotator cuff repairs were enrolled in this study. Rotator cuff tears were diagnosed by use of preoperative magnetic resonance imaging (MRI), and the size of a rotator cuff was confirmed at the time of arthroscopic operation. Indication for surgery was symptomatic full thickness rotator cuff tear or partial thickness rotator cuff more than 50% thickness in case of failed conservative therapy. Among them, 21 patients were randomly allocated into group I, and received suprascapular nerve block (SSNB) and axillary nerve block (ANB) with each 10mL ropivacaine. The other 21 patients were allocated into group II, and received SSNB with 10mL ropivacaine and ANB with 10mL normal saline.

For the cases in this study, the inclusion criteria were (1) an definite rotator cuff tear on preoperative MRI which needed repair, (2) accept an arthroscopic surgery including rotator cuff repair, (3) more than 20 years old,(4) accept preemptive regional block and patient controlled analgesia (PCA). Some patients were excluded for the following reasons (1)did not underwent arthroscopic rotator cuff repair (2) stopped PCA before postoperative 48 hours due to associated side effect (3) history of previous shoulder operation or fracture, (4) a concomitant neurologic disorder around the shoulder

Visual analogue scale (VAS) pain score, American Shoulder and Elbow Surgeons (ASES) shoulder score, Constant score, height, and weight, etc were checked preoperatively. All the regional blocks were preemptively performed under sono-guidance. PCA was set at the fixed dose (0.05 ug/kg of loading dose and 0.03ug/min.kg of continuous dose, fentanyl) to remove the effect of variable amount of PCA. VAS pain score, patient's satisfaction (SAT), the percentage of lateral pain of affected shoulder, and Lateral Pain Index (LPI: VAS × the percentage of lateral pain of shoulder ÷ 100) was checked postoperative 1, 3, 6, 12, 18, 24, 36, and 48 hours. VAS pain score was selected from 0 to 10. 0 was no pain and 10 was severe pain that the patient had ever experienced.1 SAT was also selected from 0 to 10. 0 was unsatisfactory and 10 was very satisfactory. The percentage of lateral pain was determined as a value between 0 and 100. LPI was determined as VAS pain score × the percentage of lateral pain of shoulder ÷ 100. Rebound of postoperative pain was confirmed if there had been an increase of VAS pain score after postoperative 1 hour.

Power analysis indicated that a total sample size of 34 patients (17 patients in each cohort) would provide a statistical power of 99% with a 2-sided α level of .05 to detect significant differences in VAS at postoperative 6 hours, assuming an effect size of 1.56 (mean difference: 2.5, standard deviation: 1.6). This was based on the mean and standard deviation of VAS at postoperative 6 hours observed in a pilot study of 20 patients. Double blinded randomization was performed as follows. The 48 patients who had met the inclusion criteria were randomly assigned to 1 of 2 groups depending on the combined ANB. Randomization was performed with a computer random sequence generator by an independent nurse, who prepared a syringe for combined ANB according to the assignment. The patient and all the medical staff who participated in the operation were blinded of the assignment. After this study, according to the exclusion criteria, two patient with no rotator cuff tear and three patient with only rotator cuff fraying who underwent only arthroscopic debridement were excluded from this study. One patient who stopped PCA at postoperative 1 hour was done, too. In the end, the 42 patients were included in this study. Among them, 21 patients belonged to group I, and the other 21 patients belonged to group II.

All the regional blocks were preemptively performed. When the patient was positioned in beach chair position, SSNB and ANB were performed by one anesthesiologist under sono-guidance. 23 gauge spinal needle was used. Just after skin preparation using povidone Iodine solution, a thin layer of sterile ultrasound transmission gel was placed between the ultrasound transducer and the skin. SSNB was done at first and the entry site was the mid point between an anterolateral angle of acromion and medial end of scapular spine. With the linear probe parallel to the scapular spine, the suprascapular notch was identified and the block was performed penetrating the transverse scapular ligament because the scapular nerve and artery were located at the suprascapular notch. Just after the SSNB, ANB was performed and the entry site was the point 1.5 cm medial and 2cm inferior to posterolateral angle of acromion. With the linear probe parallel to the longitudinal axis of the humerus, posterior circumflex artery was identified and the block was done at just above the artery. The color Doppler sonography may be helpful for identifying the arterial structures, but they were sometimes undetectable, and therefore they could be identified by detecting a pulsatile motion.

All the patients in this study underwent arthroscopic rotator cuff repair and subacromial decompression. All procedures were performed by one surgeon who had specialized in shoulder and elbow surgery, and sports medicine. Four routine arthroscopic portals (anterior, posterior, lateral, and posterolateral) were used in arthroscopic surgery. After bursectomy, arthroscopic subacromial decompression was performed with acromioplasty and spur removal in all patients. Suture bridge technique was mainly used for rotator cuff repair with 5.0mm Bio-Corkscrew suture anchor (Arthrex, Naples, Florida, USA) and 4.75mm Bio-SwiveLock (Arthrex, Naples, Florida, USA). Tendon to tendon suture was sometimes used for small to medium tear located around musculotendinous junction. According to the concomitant diseases, long lead of biceps (LHB) tenotomy or tenodesis, distal clavicle resection, and anterior capsulotomy were performed simultaneously.

Postoperatively, a shoulder-immobilizing sling with an abduction pillow was prescribed to each patient. The postoperative rehabilitation was individualized according to the size of rotator cuff tear and the tissue quality of torn rotator cuff. The patients without a rotator cuff tear were allowed passive forward elevation using a pulley at postoperative 48 hours just after PCA had been removed.

The normally distributed data between the groups was analyzed using a t test for independent samples. Otherwise, a nonparametric Mann-Whitney U test. Probable factors which might affect rebound of pain were analyzed using univariate logistic regression. Statistical analysis was performed using the SPSS 13.0 (SPSS Inc, Chicago, Illinois, U.S.A.). The significance level was set at P<.05.

ELIGIBILITY:
Inclusion Criteria:

1. an definite rotator cuff tear on preoperative MRI which needed repair,
2. accept an arthroscopic surgery including rotator cuff repair,
3. more than 20 years old,
4. accept preemptive regional block and PCA (patient controlled analgesia).

Exclusion Criteria:

1. did not underwent arthroscopic rotator cuff repair
2. stopped PCA before postoperative 48 hours due to associated side effect
3. history of previous shoulder operation or fracture,
4. a concomitant neurologic disorder around the shoulder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale | postoperative 48 hours
  VAS pain score was selected from 0 to 10. 0 was no pain and 10 was severe pain that the patient had ever experienced.

SECONDARY OUTCOMES:
Patient satisfaction (SAT) | postoperative 48 hours
  SAT was also selected from 0 to 10. 0 was unsatisfactory and 10 was very satisfactory.

OTHER OUTCOMES:
lateral pain index (LPI) | postoperative 48 hours
  The percentage of lateral pain was determined as a value between 0 and 100. LPI was determined as VAS pain score × the percentage of lateral pain of shoulder ÷ 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Derived] Lee JJ, Kim DY, Hwang JT, Lee SS, Hwang SM, Kim GH, Jo YG. Effect of ultrasonographically guided axillary nerve block combined with suprascapular nerve block in arthroscopic rotator cuff repair: a randomized controlled trial. Arthroscopy. 2014 Aug;30(8):906-14. doi: 10.1016/j.arthro.2014.03.014. Epub 2014 May 29. PMID 24880194